CLINICAL TRIAL: NCT01811901
Title: Reduction of In-hospital Delays in Stroke Thrombolysis: SITS-WATCH
Acronym: SITS-WATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SITS International (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20130214; 20130215
Record Dates: First submitted 2013-03-12; First posted 2013-03-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Stroke
Keywords: inhospital delays, door-to-needle time, thrombolysis, acute ischemic stroke, SITS, SITS-WATCH, stroke registry
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (SITS-WATCH centers) (Active Comparator): 15-item list of suggested interventions aiming to reduce DNT sent to SITS-WATCH centers.
  Interventions: Other: Reduction of DTN
- Control group (non SITS-WATCH centers in SITS registry) (No Intervention): Centres that do not use 15-item list of suggested interventions aiming to reduce DNT.

INTERVENTIONS:
Other: Reduction of DTN — 15-item list of suggested interventions aiming to reduce DNT sent to SITS-WATCH centers.
  Arms: Intervention group (SITS-WATCH centers)

SUMMARY:
In patients with acute ischemic stroke: the sooner the thrombolysis treatment is administered after symptom onset - the better the outcome. This delay can be dissected into onset-to-door time and door-to-needle time (DNT). SITS-WATCH aims to reduce median DNT in participating centres.

DETAILED DESCRIPTION:
In patients with acute ischemic stroke: the sooner the thrombolysis treatment is administered after symptom onset - the better the outcome. This delay can be dissected into onset-to-door time and door-to-needle time (DNT). Of the two, DNT can be directly influenced within the hospital by stream-lining of acute stroke care. The aim of our study is to reduce in-hospital delays (DNT) in self-selecting centers recruiting patients into the the Safe Implementation of Treatments in Stroke-International Stroke Thrombolysis Register (SITS-ISTR) , comprising currently more than 80 000 patients from 1338 centers. Current median of DNT in all SITS centers is 65 minutes (compared with 20 minutes in Helsinki Univer-sity Central Hospital). An itemized detailed questionnaire, including all factors known to influence DNT, has been sent to all SITS centers to identify the reasons for long in-hospital delays. Based on the replies, we have prepared a list of interventions that can be considered by individual SITS centers in order to reduce DNT with interventions that are in line with national legislation.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with acute ischemic stroke registered in SITS registry.

Exclusion Criteria:

* Centers not inputing patient data into SITS registry. Patients with missing DNT data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Absolute DNT reduction of at least 20 minutes or at least 20% change in SITS-WATCH centers that completed the whole study period | January 2013-December 2014
  DNT will be evaluated at regular intervals (twice a year).

SECONDARY OUTCOMES:
Significantly larger reduction of DNT in SITS-WATCH centers compared with non-SITS-WATCH centers in SITS. | 2014-2015
  Proportion of centers with median DNT below 40 minutes. At least 3 new interventions implemented. Percentage of implemented interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- SITS International / Karolinska Hospital, Stockholm, Sweden